CLINICAL TRIAL: NCT00222742
Title: Pediatric Traumatic Brain Injury Consortium: Hypothermia
Brief Title: Hypothermia in Children After Trauma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Phoenix Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01-NS052478-01; 1R01NS052478-01
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Traumatic Brain Injury
Keywords: hypothermia; pediatric TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypothermia | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Induced moderate hypothermia (32-33 C)
  Interventions: Procedure: induced moderate hypothermia

INTERVENTIONS:
Procedure: induced moderate hypothermia — Subjects assigned to the treatment arm will be cooled to 32-33 °C for 48 hours and then slowly warmed.

SUMMARY:
The primary hypothesis for this application for a multicenter phase III randomized clinical trial (RCT) is that induced moderate hypothermia (HYPO) (32-33 °C) after severe traumatic brain injury (TBI) in children and maintained for 48 hours will improve mortality at 3 months and 12 month functional outcome as assessed by the Glasgow Outcome Scale (GOS).

DETAILED DESCRIPTION:
The primary specific aim of this RCT is to determine the effect of induced moderate HYPO (32-33 °C) after severe TBI in children on mortality at 3 months post injury. The primary outcome measure will be the GOS; the primary time point for evaluation is 3 months. Further secondary functional outcome measures will include the GOS - Extended Pediatrics (GOS - E Peds), and Vineland Adaptive Behavior Scale (VABS) and will be assessed in conjunction with the GOS at 6 and 12 months post injury.

The secondary hypotheses are based on the results and analysis of the Pilot Clinical Trial (completed and recently published [Adelson et al. NEUROSURGERY. 56 (4): 740-754, 2005]). These secondary hypotheses include that induced moderate hypothermia (HYPO) (32-33 °C) after severe TBI in children and maintained for 48 h:

* will improve other outcome assessments including neurocognitive status on performance-based neuropsychological testing across the domains of intellectual development, learning and memory, language, motor and psychomotor skills, visuo-spatial abilities, attention and executive function, and behavior at only 6 and 12 months after injury;
* HYPO will improve long term outcome of all age ranges and across genders in infants, young, preadolescent, and adolescent children; AND
* HYPO will lessen intracranial hypertension and lessen the intensity of therapy necessary for control of ICP.

Based on these hypotheses, further secondary specific aims are proposed:

* Specific Aim 2: To determine the effect of early induced moderate HYPO (32-33°C) after severe TBI in children on global function and neurocognitive outcomes in the areas of intellectual ability/ development, memory and learning, and behavior at 6 and 12 months post injury.
* Specific Aim 3: To determine the effect of early induced moderate HYPO after severe TBI in children of different age ranges (< 6 y and 6- < 16 y) on mortality and 6 and 12 months functional and neurocognitive outcomes.
* Specific Aim 4: To determine the effect of early moderate HYPO after severe TBI in children on reducing intracranial hypertension and maintaining adequate cerebral perfusion pressure (CPP).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a GCS </= 8
2. Glasgow Motor Score < 6
3. Closed head injury
4. Age 0 < 18 y

Exclusion Criteria

1. Unavailable to initiate cooling within 6 hours of injury
2. Glasgow Coma Scale (GCS) score = 3 and abnormal brainstem function
3. Normal initial CT scan (No blood, fracture, swelling, and/or shift)
4. Penetrating brain injury
5. No known mechanism of injury
6. Unknown time of injury
7. Uncorrectable coagulopathy (PT/PTT > 16/40 sec, INR > 1.7)
8. Hypotensive episode (Systolic Blood Pressure <5th percentile for age>10 min)
9. Documented Hypoxic episode (O2 saturation < 94% for > 30 min)
10. Pregnancy

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2007-11; Primary Completion 2011-05 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary specific aim of this RCT is to determine the effect of induced moderate HYPO (32-33 °C) after severe TBI in children on mortality. | 3 month post injury

SECONDARY OUTCOMES:
To determine the effect of HYPO after severe TBI in children on global function and neurocognitive outcomes in the areas of intellectual ability/development, memory and learning, and behavior. | at 6 and 12 months post injury
To determine the effect of HYPO after severe TBI in children of different age ranges (< 6y; 6-<16y; and 16-<18y) on mortality and 6 and 12 months functional and neurocognitive outcomes. | 3, 6 and 12 months post injury
To determine the effect of HYPO after severe TBI in children on reducing intracranial hypertension and maintaining adequate cerebral perfusion pressure (CPP). | 7 days post injury

CONTACTS AND LOCATIONS:
Overall Officials: P. David Adelson, MD, Principal Investigator — Phoenix Children's Hospital
Locations (30):
- United States (17):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of California, Davis Medical Center, Sacramento, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Cohen's Children's Hospital, New Hyde Park, New York
  - Weill Cornell Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh/Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington
- Australia (7):
  - Sydney Children's Hospital, Randwick, Sydney, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Brisbane, Queensland
  - Mater Children's Hospital, Brisbane, Queensland
  - Children's Youth and Women's Health Service, North Adelaide, South Australia
  - Royal Children's Hospital Melbourne, Parkville, Victoria
  - Princess Margaret Hospital for Children, Subiaco, Perth, Western Australia
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
- Starship Children's Hospital, Auckland, New Zealand
- University of Cape Town, Rondebosch, Cape Town, South Africa
- United Kingdom (2):
  - Institute of Child Health, Univ. College London & Great Ormond, Bloomsbury, London
  - Birmingham Children's Hospital, Birmingham, West Midlands

REFERENCES:
- [Derived] Meinert E, Bell MJ, Buttram S, Kochanek PM, Balasubramani GK, Wisniewski SR, Adelson PD; Pediatric Traumatic Brain Injury Consortium: Hypothermia Investigators. Initiating Nutritional Support Before 72 Hours Is Associated With Favorable Outcome After Severe Traumatic Brain Injury in Children: A Secondary Analysis of a Randomized, Controlled Trial of Therapeutic Hypothermia. Pediatr Crit Care Med. 2018 Apr;19(4):345-352. doi: 10.1097/PCC.0000000000001471. PMID 29370008
- [Derived] Adelson PD, Wisniewski SR, Beca J, Brown SD, Bell M, Muizelaar JP, Okada P, Beers SR, Balasubramani GK, Hirtz D; Paediatric Traumatic Brain Injury Consortium. Comparison of hypothermia and normothermia after severe traumatic brain injury in children (Cool Kids): a phase 3, randomised controlled trial. Lancet Neurol. 2013 Jun;12(6):546-53. doi: 10.1016/S1474-4422(13)70077-2. Epub 2013 May 8. PMID 23664370